CLINICAL TRIAL: NCT01239251
Title: Feasibility of Using the GlowCap Reminder System in Patients With Early Stage Breast Cancer Receiving Adjuvant Endocrine Therapy
Brief Title: GlowCap Reminder System in Patients With Early Stage Breast Cancer Receiving Adjuvant Endocrine Therapy
Status: Terminated | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 10-183
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: GlowCap; adjuvant endocrine therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- breast cancer patients taking endocrine therapy: Breast cancer patients, currently taking adjuvant endocrine therapy will be equipped with a GlowCap device for a period of 30 days. The GlowCap will become part of their medication taking routine.
  Interventions: Other: GlowCap device

INTERVENTIONS:
Other: GlowCap device — Participants will be provided with a device called the GlowCap for a period of 30 days. The device has visual and auditory cues to help patients remember to take their medication at the same time each day. The GlowCap will be programmed to glow when it is time for each patient to take her medication. The GlowCap will initially glow bright orange for the first hour from the time the patient is scheduled to take the medication. During the second hour, the GlowCap system will play music in addition to continuing to glow. If after 2 hours the patient still has not opened the medication bottle, she will receive a phone call reminding her to take her medication.

SUMMARY:
The purpose of this study is to test the ease of using a new device, called the GlowCap that reminds the patient to take their breast cancer hormone pill. The study will collect information about the experience with this device and what the patient thinks of its role in the daily pill taking routine.

ELIGIBILITY:
Inclusion Criteria:

* Early stage breast cancer patients taking adjuvant endocrine therapy (ie, tamoxifen, anastrozole, letrozole, exemestane).
* Age ≥ 60 years
* Must have broadband internet access at home (to enable the base for the system to communicate to the Vitality server).
* Must have a landline or mobile phone

Exclusion Criteria:

* Non-English speaking patients

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast Cancer Medicine practice outpatients
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Assess the usability of the GlowCap system by patients | 2 years
  >60 years of age with early stage breast cancer.

SECONDARY OUTCOMES:
Measure the acceptance and satisfaction of the GlowCap reminder system | 2 years
  with respect to medication adherence in patients >60 years with early stage breast cancer taking adjuvant endocrine therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Traina, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center 1275 York Avenue, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm